CLINICAL TRIAL: NCT07011238
Title: Alloreactive Memory B Lymphocytes and Anti-HLA Sensitization in Kidney Transplantation
Brief Title: Alloreactive Memory B Lymphocytes and Anti-HLA Sensitization
Acronym: ALLO-BMEM
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/301/OB; 2021-A02507-34 (Other: ANSM)
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Kidney Transplant
Keywords: B lymphocytes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — volume 50 ml of whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Patients meeting HLA immunization criteria — At enrollment visit, a single sample of a volume of 50 ml of blood will be taken as part of routine care in order to directly and simultaneously explore the clonality (BCR repertoire), the phenotype of membrane markers and the transcriptome of Bmem alloreactive with respect to a restricted panel of HLA alleles chosen according to the HLA antibody reactivity profile of the patients analyzed

SUMMARY:
In transplantation, B lymphocytes are major cellular players in the alloreactive humoral response through the production of antibodies targeting allogeneic HLA molecules expressed by the transplant. In subjects sensitized to HLA antigens, the contribution of pre-existing alloreactive memory B lymphocytes (Bmem) to allograft rejection phenomena after transplantation is now recognized. It has been proposed that the identification of these Bmem during the pre-transplant period could contribute to a better assessment of post-transplant immunological risk, allowing optimization of strategies to prevent humoral rejection. However, knowledge regarding the phenotypic and functional heterogeneity of Bmem as well as their clonal diversity is still extremely limited, not allowing discrimination between pathogenic and non-pathogenic alloreactive humoral responses. Such discrimination requires a better understanding of the modalities of differentiation of alloreactive B lymphocyte responses. To this end, this study aims to characterize the clonal, phenotypic and functional properties of alloreactive Bmem in subjects awaiting renal transplantation and sensitized to HLA antigens.

DETAILED DESCRIPTION:
The hypothesis of this study is that analyzing the heterogeneity of alloreactive Bmem in patients carrying HLA antibodies under varying HLA immunization intensity conditions (corresponding to varying intensities of exposure to HLA alloantigens) is likely to provide insight into the differential modalities of overall alloreactive B repertoire formation.

Two types of patients sensitized to HLA antigens following immunizing events (at least one transplant or pregnancy) awaiting kidney transplantation will be specifically explored:

* patients deemed hyperimmunized based on an incompatible graft rate (IGR) ≥ 85%, carrying a broad HLA antibody repertoire
* patients immunized with an IGR between 50 and 85%, carrying a more restricted HLA antibody repertoire. These two groups will be characterized by differential intensities of exposure to HLA alloantigens. Patients with a history of immunizing events other than transfusions will not be investigated, due to the lack of detection of alloreactive Bmem in this situation.

"Control" patients will also be included: "naïve" patients carrying HLA antibodies in the absence of a classic immunizing event, in whom alloreactive Bmem are not detectable.

The exploration of alloreactive Bmem in these two groups aims to identify potential differences in terms of clonality, phenotype, and functionality, which could clarify several aspects of the alloreactive humoral response:

The expected impact of this pilot translational study in kidney transplantation is threefold:

* the acquisition of fundamental knowledge in the field of alloantigen-specific human Bmem biology
* the acquisition of data prior to the subsequent exploration of the characteristics of the alloreactive B cell response during acute or chronic humoral rejection
* and ultimately, the identification of phenotypic, clonotypic, or functional markers that could potentially be used to better discriminate the immunological risk associated with the presence of antibodies and HLA-reactive B cells.

The low frequency of alloreactive Bmem, estimated at 20-150 per million B lymphocytes (for a given HLA specificity), as well as the number and epitopic diversity of targeted HLA antigens, complicate the direct assessment of their repertoire and functionalities. High-throughput approaches (RNAseq) in single cells, which have become essential for characterizing the heterogeneity of rare cellular contingents, now make it possible to simultaneously interrogate the repertoire and transcriptome of immune cells. In this project, we will take advantage of these recent methodologies to directly and simultaneously explore the clonality (BCR repertoire), the phenotype of membrane markers and the transcriptome of alloreactive Bmem towards a restricted panel of HLA alleles chosen according to the HLA antibody reactivity profile of the patients analyzed. This methodology allows the acquisition of individual characteristics of several hundred alloreactive B lymphocytes per patient and their comparison with polyclonal Bmem from patients or control subjects. This is a pilot study intended to acquire preliminary data prior to studies on a larger number of patients, before and after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Rouen University Hospital patient monitored in the Nephrology and Kidney Transplantation Department, registered on the national kidney transplant waiting list
* Carrier of HLA antibodies, including at least anti-HLA2, identified during the last screening
* Notion of classic immune-promoting events including at least one previous transplant or pregnancy, or absence of a known immune-promoting event (naïve patient group)
* Incompatible graft rate (IGR)

  * IGR ≥ 85% (hyperimmunized patient group with anti-HLA polyreactivity) or
  * IGR between 50% and 85% (immunized patient group with a more restricted repertoire of HLA reactivities) or
  * IGR < 50% (naïve patient group with no known history of immune-promoting events)
* Person who has read and understood the information letter and does not object Not participating in the study
* Affiliation to a social security scheme

Exclusion Criteria:

* Patients who have received rituximab in the previous year (B-cell depleting therapy)
* Patients undergoing an HLA desensitization protocol using plasmapheresis and/or rituximab
* Patients with an active infection
* Persons deprived of their liberty by an administrative or judicial decision or persons placed under judicial protection/guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients awaiting kidney transplantation and carrying HLA antibodies following immunizing events
Sampling Method: Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-04-17 (Estimated); Study Completion 2026-05-17 (Estimated)

PRIMARY OUTCOMES:
Level of heterogeneity of alloreactive Bmem targeting HLA alloantigens | At enrollment visit
  The main objective is to determine the level of heterogeneity of alloreactive Bmem targeting HLA alloantigens of given specificities (primarily HLA-A2) in patients awaiting kidney transplantation and carrying HLA antibodies following immunizing events by evaluating the number of alloreactive Bmem clusters identified (in all patients) on the basis of their gene expression profiles (bioinformatics analysis of expression data with the open source Seurat suite

SECONDARY OUTCOMES:
Evaluation of the level of phenotypic heterogeneity of alloreactive Bmem | At enrollment visit
  To compare the level of phenotypic heterogeneity of alloreactive Bmem of given specificities (including HLA-A2) according to the immunization profile (hyperimmunization versus more restricted immunization) by evaluating the number of alloreactive Bmem clusters identified (in all patients) on the basis of their gene expression profiles (bioinformatics analysis of expression data with the open source Seurat suite
Evaluation of the level of transcriptional heterogeneity of alloreactive Bmem | At enrollment visit
  To compare the level of transcriptional heterogeneity of alloreactive Bmem of given specificities (including HLA-A2) according to the immunization profile (hyperimmunization versus more restricted immunization) by evaluating the number of alloreactive Bmem clusters identified (in all patients) on the basis of their gene expression profiles (bioinformatics analysis of expression data with the open source Seurat suite
Clonality of Bmem specific to each HLA antigen tested | At enrollment visit
  Evaluation of VDJ junction sequences of IgH genes coding for the BCR of alloreactive Bmem, analyzed with the IgBlast tool
Somatic mutations of the BCR of Bmem IgG+ or IgM+ | At enrollment visit
  Determine the number of somatic mutations of the BCR of Bmem IgG+ or IgM+ in each patient, and according to the IgBlast immunization profile (calculation of the average number of somatic mutations of the VDJ junction of the IgH genes)
Ratio of the number of Bmem IgM+/IgG+ | At enrollment visit
  Determination of the Bmem IgM+/IgG+ ratio in each patient based on the immunization profile

CONTACTS AND LOCATIONS:
Locations (1):
- University Hopsital of Rouen, Rouen, France

IPD SHARING:
Plan to Share IPD: Yes
The data provided will be the property of the sponsor and will be used solely for its own research activities.